CLINICAL TRIAL: NCT04340830
Title: The Effect of Smoking on Dimensional Changes of Free Gingival Graft Around Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Oya Turkoglu, Professor, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-DIS-011
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Smoking; Free Gingival Graft; Dental Implant
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smoker (Experimental): Those consuming at least 10 cigarette a day for ten years were included in smoker group.
  Interventions: Procedure: Free gingival graft
- non-smoker (Active Comparator): Patients who never smoke were included in non-smoker group. Patients who quit smoking were not included in this group.
  Interventions: Procedure: Free gingival graft

INTERVENTIONS:
Procedure: Free gingival graft — Following recipient site preparation, free gingival graft obtained from palatal mucosa was applied to buccal sites of dental implants having inadequate keratinized attached mucosa.

SUMMARY:
There are studies investigating the dimensional changes following free gingival graft (FGG) around teeth with inadequate attached gingiva, however no study investigating the effect of smoking on dimensional changes following FGG around dental implants exists. In the present study, we hypothesized that smoking might increase the dimensional change of FGG around dental implants and affect the healing of donor site.

ELIGIBILITY:
Inclusion Criteria:

Implants with inadequate attached gingiva on the buccal site, which placed in posterior region at least 1 year ago, and loaded with a fixed prosthetic restoration at least 6 months ago.

Exclusion Criteria:

Implants with peri-implantitis, patients who had previously the soft or hard tissue graft surgery at the site in question, patients who had previously operated from the donor site, patients with systemic disease that may interfere with periodontal surgery, patients taking any medication that can prolong bleeding, patients with immune system disease, infectious diseases such as hepatitis or HIV, individuals under the age of 18, and women with pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
dimensional change of free gingival graft | 0,1, 3, 6 months
  the changes in vertical dimension of free gingival graft was measured by functional and visual methods intra-orally by individual stents, and horizontal dimension of free gingival graft was measured on digital photographs using specific software.
change in total free gingival graft area | 0, 7th day, 1,3, 6 months
  total free gingival graft area was calculated on digital photographs using specific software.

SECONDARY OUTCOMES:
Depth of vestibule sulcus | 0, 7th day, 1,3, 6 months
tissue thickness of recipient and donor sites | 0, 7th day, 1,3, 6 months
VAS | 0,1,2,3,4,5,6,7. days